CLINICAL TRIAL: NCT06905886
Title: Impact of Menopausal Hormone Therapy on Resting Energy Expenditure in Postmenopausal Women
Brief Title: Resting Energy Expenditure in Postmenopausal Women
Acronym: MenoBOLISM
Status: Not yet recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-01570
Record Dates: First submitted 2025-03-31; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Postmenopause; Energy Expenditure; Hormone Replacement Therapy

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Biospecimen Retention: Samples Without DNA — Blood samples - serum / plasma, to assess hormone concentrations (e.g., estradiol, progesterone, LH, FSH). Serum / plasma does not contain DNA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Menopausal Hormone Therapy (MHT): Postmenopausal women, receiving Menopausal Hormone Therapy for 4 weeks, following an observation phase of 2 weeks without intervention.

SUMMARY:
Obesity and its associated comorbidities are rising at an alarming rate, particularly among postmenopausal women. Menopause, characterized by a decline in estradiol and progesterone levels, is often accompanied by weight gain. Fear of this weight gain is a major reason why many women hesitate to initiate or continue menopausal hormone therapy (MHT), with discontinuation often occurring within the first few months. However, scientific evidence on whether MHT influences weight gain remains inconclusive. A Cochrane Review found no significant effect of estrogen or combined estrogen-progestogen therapy on menopause-related weight gain, suggesting that aging and lifestyle changes play a more prominent role.

While the effects of estrogen on energy intake have been well-documented, data on its impact on energy expenditure-particularly resting energy expenditure (REE), the largest component of total energy expenditure-are scarce. Several studies suggest that sex hormones may influence REE, as observed in premenopausal women, where REE increases during the luteal phase when estradiol and progesterone levels are high. However, findings on this topic remain inconsistent, and it is unclear whether estrogen or progesterone plays the primary role. Research on the effects of exogenous hormone administration, such as MHT, on REE is extremely limited, with existing studies producing mixed results. Additionally, the potential influence of progestogens on REE has been largely overlooked. Given that a low REE is a strong predictor of weight gain and obesity, understanding the effects of MHT on REE is crucial.

This observational clinical trial aims to investigate the precise effect of MHT (estradiol + progesterone) on REE in postmenopausal women with an indication for MHT. Secondary objectives include examining MHT's impact on energy intake, physical activity energy expenditure, performance capacity, body composition, core body temperature, serum hormone profiles (luteinizing hormone, follicle-stimulating hormone, estradiol, progesterone), glucose metabolism, fasting blood lipid levels, and miRNA expression (miR-370 and miR-29b, which are involved in lipid and glucose metabolism). Additionally, the study will assess various aspects of subjective well-being and quality of life.

By addressing the current gaps in scientific knowledge, this study seeks to provide robust evidence on the role of MHT in energy metabolism, potentially reshaping perspectives on its risks and benefits in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Healthy postmenopausal woman
* Indication for MHT (e.g. climacteric syndrome, osteoporosis, etc.)
* Body Mass Index (BMI) 18.5 - 29.9 kg/m2
* Non smoker
* Willingness to maintain unchanged dietary habits and the type and frequency of sports activities throughout the entire 6-week study period. I.e. no dietary changes/restrictions, start of a special exercise program or start of any weight-loss measures are planned during the study period.

Exclusion Criteria:

* Pregnancy or Lactation
* Other clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease, etc.)
* Systemic hormone therapy or hormonal contraception (estrogens, progestogens, androgens) during the study and within 12 weeks prior to study entry
* Phytotherapeutics for therapy of climacteric syndrome during the study and within 12 weeks prior to study entry
* Use of psychotropic drugs and other drugs that have an influence on resting energy expenditure during the study and within 12 weeks prior to study entry
* Substance abuse (e.g. nicotine, alcohol, drugs)
* Use of appetite suppressants
* Hypersensitivity or allergy to class of drugs or to any ingredients of the used IMPs (Oestrogel® and Utrogestan®)
* Contraindication for estradiol or progesterone medication according to swissmedicinfo.ch: Neoplasia of the breast or other sexual organ; Benign or malignant liver tumors; Acute or chronic liver disease; Cholestatic jaundice; Porphyria; Arterial or venous thromboembolic events; Abnormal genital bleeding of unknown cause
* Use of medication with active ingredients that interact with the metabolization of estradiol or progesterone. For each medication a drug interaction check will be performed: Lexicomp® Drug Interactions, UpToDate®
* Known or suspected non-compliance due to inability to follow the procedures of the study (e.g. illiteracy, language problems, psychological disorders, dementia, etc.)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postmenopausal women with an indication for MHT (e.g. climacteric syndrome, osteoporosis, etc.). Women will be recruited at the University Hospital of Bern, Switzerland - Department of Gynecological Endocrinology and Reproductive Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Resting Energy Expenditure (REE) | 4 weeks
  Difference in absolute REE (kcal/day) before hormonal substitution and after four weeks of MHT

CONTACTS AND LOCATIONS:
Overall Officials: Susanna Weidlinger, Dr. med., Principal Investigator — Department of Gynecologic Endocrinology and Reproductive Medicine, University Clinic for Gynecology, University Hospital Bern
Locations (1):
- University Hospital of Bern, Switzerland; Department of Gynecological Endocrinology and Reproductive Medicine, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No
Because IPD contain health-related data.